CLINICAL TRIAL: NCT06112392
Title: Stellate Ganglion Block in Patients With Advanced Primary Parkinson's Disease: a Small, Open, Randomized Controlled Clinical Study
Brief Title: Clinical Study of Stellate Ganglion Block in Treatment of Patients With Advanced Primary Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Gao Xiaoya, Chief Physician, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-KY-080-01
Record Dates: First submitted 2023-07-13; First posted 2023-11-01 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Stellate Ganglion; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's disease group (Experimental): Diagnostic criteria: Patients with Parkinson's disease who met the diagnostic criteria for MDS as "probable PD" or" confirmed PD" in 2016
  Inclusion criteria:
  1. Age 40-85;
  2. Patients with Parkinson's disease who met the diagnostic criteria of MDS as "probable PD" or" confirmed PD" in 2016;
  3. The patient or his/her legal guardian agrees to participate in the study and signs the informed consent;
  4. Hoehn-yahr (H&Y) 3 ~ 5;
  Interventions: Diagnostic Test: Treatment （Stellate ganglion block；Oral standard anti-Parkinson's drugs）
- Non-parkinson's disease group (Experimental): Exclusion criteria:
  1. Allergic to local anesthetic drugs;
  2. Unable to cooperate with motor or non-motor function monitoring;
  3. Patients with Parkinson's superposition syndrome, such as cortical basal ganglia degeneration, lewy body dementia, multisystem atrophy and progressive supranuclear palsy, were excluded; Patients with secondary Parkinson's disease, such as vascular Parkinson's disease, drug toxicity or traumatic Parkinson's disease;
  4. Refuse to sign the consent form.
  Interventions: Diagnostic Test: Treatment （Oral standard anti-Parkinson's drugs）

INTERVENTIONS:
Diagnostic Test: Treatment （Stellate ganglion block；Oral standard anti-Parkinson's drugs） — Treatment （Stellate ganglion block；Oral standard anti-Parkinson's drugs）
  Arms: Parkinson's disease group
Diagnostic Test: Treatment （Oral standard anti-Parkinson's drugs） — Treatment （Oral standard anti-Parkinson's drugs）
  Arms: Non-parkinson's disease group

SUMMARY:
At present, there are no reports on the application of stellate ganglion block in the treatment of Parkinson's disease patients at home and abroad. Based on the preliminary clinical observation, this project intends to apply stellate ganglion block in the treatment of patients with intermediate and advanced Parkinson's disease through an open, randomized controlled small sample clinical study. To determine whether stellate ganglion block can effectively improve motor symptoms and non-motor symptoms in patients with primary advanced Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a relatively common degenerative disease of the central nervous system. In the past few decades, China's population has increased significantly, resulting in a rapid increase in the number of elderly people. According to the 2016 Global Burden of Disease study, the number of PD patients in China accounts for about 23% of the global PD population. By the end of 2020, the estimated number of people living with Parkinson's disease in China is about 3.62 million, and it is expected that by 2030, 50% of the world's PD patients will be Chinese. The main manifestations of Parkinson's disease are motor symptoms such as bradykinesia, myotonia and tremor, and non-motor symptoms such as autonomic nervous dysfunction, sleep disturbance and anosmia.

Both motor symptoms and non-motor symptoms can significantly affect patients' quality of life. At present, the domestic and foreign treatment guidelines for Parkinson's disease still prefer drug therapy represented by dopa. However, in the middle and late stages of the disease, side effects such as symptom fluctuation or hyperactivity disorder complicated by long-term drug use gradually appear, and the efficacy of patients on levodopa declines, which seriously affects the quality of life of patients. For patients with advanced Parkinson's disease, current anti-Parkinson's guidelines advocate a combination of drug therapy and non-drug therapy. As a major non-drug treatment for Parkinson's disease, deep brain stimulation (DBS) has limited its wide clinical application due to its complex, invasive, expensive, and many side effects, while conventional rehabilitation therapy is limited to functional exercise such as speech and swallowing, with limited efficacy. Therefore, the search for new treatments for Parkinson's disease is imperative.

At present, there are no reports about the application of SGB in the treatment of patients with Parkinson's disease at home and abroad. Based on the preliminary clinical observation, this study intends to apply SGB in the treatment of patients with advanced Parkinson's disease through an open, randomized controlled small sample clinical study, so as to confirm that SGB can effectively improve the motor symptoms and non-motor symptoms of patients with advanced Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease who met the diagnostic criteria for MDS as "probable PD" or" confirmed PD" in 2016

Inclusion criteria:

1. Age 40-85;
2. Patients with Parkinson's disease who met the diagnostic criteria of MDS as "probable PD" or" confirmed PD" in 2016;
3. The patient or his/her legal guardian agrees to participate in the study and signs the informed consent;
4. Hoehn-yahr (H&Y) 2.5 ~ 5;

Exclusion Criteria:

* 1. Allergic to local anesthetic drugs;

  2. Unable to cooperate with motor or non-motor function monitoring;

  3. Patients with Parkinson's superposition syndrome, such as cortical basal ganglia degeneration, lewy body dementia, multisystem atrophy and progressive supranuclear palsy, were excluded; Patients with secondary Parkinson's disease, such as vascular Parkinson's disease, drug toxicity or traumatic Parkinson's disease;

  4. Refuse to sign the consent form.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Improved MDS-UPDRS scale scoring | 12 weeks
  The revised Movement Disorders Association Unified Parkinson's Disease Rating Scale has four major components, all of which include both physician and patient aspects. The first component is psychological, behavioral and emotional. The second part is daily life activities; The third part is motor symptoms; The fourth part is complications.

SECONDARY OUTCOMES:
NMSS (Non-motor Symptom Evaluation Scale) | 12 weeks
  Non-motor Symptom Evaluation Scale, minimum value 0 points, maximum 360 points. The higher the score, the worse the condition.
Pdq-39 (Self-rating Scale for clinical evaluation of quality of life in patients with Kinson disease) | 12 weeks
  Self-rating Scale for clinical evaluation of quality of life in patients with Kinson disease, minimum value 0 points, maximum 156 points. The higher the score, the worse the condition.
H&Y classification (Classification of Parkinson's disease) | 12 weeks
  Classification of Parkinson's disease, minimum value 0 points, maximum 5 points. The higher the score, the worse the condition.
LDE (Levodopa Equivalent dose) | 12 weeks
  Levodopa Equivalent dose, based on the dose of different anti-Parkinson's drugs. The higher the score, the worse the condition.
Hamilton Anxiety Scale (HAMA) | 12 weeks
  Hamilton Anxiety Scale, minimum value 0 points, maximum 56 points. The higher the score, the worse the condition.
Parkinson's Disease Sleep Scale (PDSS) | 12 weeks
  Parkinson's Disease Sleep Scale, minimum value 0 points, maximum 150 points. The higher the score, the better the patient.
Montreal Cognitive Assessment Scale | 12 weeks
  Montreal Cognitive Assessment Scale, minimum value 0 points, maximum 30 points. The higher the score, the better the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoya Gao, doctor, Principal Investigator — Southern Medical University, China
Locations (1):
- Zhujiang Hospiatal, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Qi S, Yin P, Wang L, Qu M, Kan GL, Zhang H, Zhang Q, Xiao Y, Deng Y, Dong Z, Shi Y, Meng J, Chan P, Wang Z. Prevalence of Parkinson's Disease: A Community-Based Study in China. Mov Disord. 2021 Dec;36(12):2940-2944. doi: 10.1002/mds.28762. Epub 2021 Aug 14. PMID 34390510
- [Result] Santos-Garcia D, de la Fuente-Fernandez R. Impact of non-motor symptoms on health-related and perceived quality of life in Parkinson's disease. J Neurol Sci. 2013 Sep 15;332(1-2):136-40. doi: 10.1016/j.jns.2013.07.005. Epub 2013 Jul 25. PMID 23890935
- [Result] Jost WH, Buhmann C. The challenge of pain in the pharmacological management of Parkinson's disease. Expert Opin Pharmacother. 2019 Oct;20(15):1847-1854. doi: 10.1080/14656566.2019.1639672. Epub 2019 Jul 10. PMID 31290336
- [Result] Stozek J, Rudzinska M, Pustulka-Piwnik U, Szczudlik A. The effect of the rehabilitation program on balance, gait, physical performance and trunk rotation in Parkinson's disease. Aging Clin Exp Res. 2016 Dec;28(6):1169-1177. doi: 10.1007/s40520-015-0506-1. Epub 2015 Dec 10. PMID 26661467
- [Result] Bi Y, Wang B, Yin Z, Zhang G, Chen H, Wang M. [Effects of stellate ganglion block on AMP-ativated protein kinase and astrocyte in hippocampal neurons in postoperative aged rats]. Zhonghua Yi Xue Za Zhi. 2014 Jul 22;94(28):2222-6. Chinese. PMID 25331477
- [Result] Dai D, Zheng B, Yu Z, Lin S, Tang Y, Chen M, Ke P, Zheng C, Chen Y, Wu X. Right stellate ganglion block improves learning and memory dysfunction and hippocampal injury in rats with sleep deprivation. BMC Anesthesiol. 2021 Nov 8;21(1):272. doi: 10.1186/s12871-021-01486-4. PMID 34749669
- [Result] Uchida K, Tateda T, Hino H. Novel mechanism of action hypothesized for stellate ganglion block related to melatonin. Med Hypotheses. 2002 Oct;59(4):446-9. doi: 10.1016/s0306-9877(02)00158-5. PMID 12208186
- [Result] Moon HS, Chon JY, Lee SH, Ju YM, Sung CH. Long-term Results of Stellate Ganglion Block in Patients with Olfactory Dysfunction. Korean J Pain. 2013 Jan;26(1):57-61. doi: 10.3344/kjp.2013.26.1.57. Epub 2013 Jan 4. PMID 23342209

DOCUMENTS (2):
  • Study Protocol (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT06112392/Prot_000.pdf
  • Informed Consent Form (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT06112392/ICF_001.pdf